CLINICAL TRIAL: NCT04039438
Title: Relationships Among Interest and Importance of Activities, Sedentary Behaviors, and Socio-demographic Factors in Sedentary Older Adults in the Community
Brief Title: Relationships Among Sedentary Behaviors and Other Factors
Status: Completed | Type: Observational
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Young Joo Kim, Assistant Professor, East Carolina University
Other Study IDs: UMCIRB 19-001417
Record Dates: First submitted 2019-07-24; First posted 2019-07-31 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Older Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention will be provided during the study nor participants will be receiving any intervention anywhere else.

SUMMARY:
Due to the increasing sedentary behaviors in older adults, it is important to understand the factors related to sedentary behaviors. Although systematic reviews have identified sociodemographic and environmental factors related sedentary behaviors, no study on the relationships between interested and important activities and sedentary behaviors in older adults was found.

In this study, investigators aim to investigate the relationships among interested and important activities, sedentary behaviors, and sociodemographic factors in older adults living in the community. Investigators will recruit 30 sedentary older adults living in the community who are cognitively intact, have no physical limitations, and are medically stable. Participants will be assessed once using subjective and objective measures:

1) estimated energy expenditure levels for interested, important, and current activities, 2) time spent on sedentary activities, and 3) sociodemographic factors.

The results of this study will provide supporting evidence for the role of meaningful occupations to decrease sedentary behaviors. In addition, the results may show the relevant sociodemographic factors that occupational therapy practitioners need to be aware when encouraging active lifestyle for sedentary older adults in the community.

ELIGIBILITY:
Inclusion Criteria:

* age of 65 years or older
* intact cognition confirmed by the Montreal Cognitive Assessment Blind score 18 or greater
* self-report of no physical activity restrictions from the physician
* sedentary lifestyle confirmed by the Rapid Assessment Disuse Index score 26 or greater,
* living 30 miles from the College of Allied Health Sciences at East Carolina University

Exclusion Criteria:

* An acute or terminal illness
* a myocardial infarction in the past 6 months
* unstable cardiovascular or metabolic disease
* neuromusculoskeletal disorders severely disrupting voluntary movement
* limb amputation
* upper or lower extremity fracture in the past 3 months
* current symptomatic hernias or hemorrhoids
* cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Medically stable older adults
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Activity Card Sort | One time during the initial, one-time study visit about their current stauts (participants are visited only once in the study)
  The Activity Card Sort assesses the participation level in instrumental, leisure, and social activities. The Activity Card Sort uses 89 photographs. For each photograph, participants will be asked if they are interested in doing the activity in each photograph, if the activity in each photograph is important for them to do, and if participants are currently doing it. Then, Three mean metabolic equivalent levels of interested, important, and current activities will be calculated.
Physical activity level | 10-14 consecutive days, 24/hours a day, following the initial, one-time visit (participants are visited only once in the study)
  Physical activity level measured by ActiGraph GT9X Link. The data will be collected for at least 7-full days to record the pattern of activity levels of a week.
Sociodemographic form | One time during the initial, one-time study visit about their current status (participants are visited only once in the study)
  The information will be used to determine the characteristics of the participants and generalizability of the results, and to determine the relationships with interested, important, and current activities. The form collects socio-demographic information, such as race, gender, highest education received, living status, occupations, total household annual income, recent hospitalization, cardiovascular risk factors, the number of medications taken daily, and weekly exercise level. Information is all self-reported.

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No